CLINICAL TRIAL: NCT01493128
Title: Ultrastructure of Sarcolemma, Immunofluorescence of Calcium Handling Proteins and Mitochondrial Function in Atrial Myocytes of Patients in Sinus Rhythm and With Atrial Fibrillation
Brief Title: Ultrastructure of Atrial Myocytes in Patients in Sinus Rhythm and With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ABJ01
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial cells; myocardial tissue; t-tubules; immunofluorescence
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Myocardial tissue from the right and left atrial appendage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- stable sinus rhythm
- permanent atrial fibrillation
- paroxysmal atrial fibrillation

SUMMARY:
The aim of this work is to study the prevalence of T-tubular system in left and right myocytes from patients in sinus rhythm and whether this is altered in paroxysmal and permanent atrial fibrillation. Furthermore, since current information is lacking on the key Ca2+-handling proteins RyR, NCX, and SERCA-2a from patients in Atrial Fibrillation (AF), it will be investigated whether a regulation of these proteins could be an underlying cause of the disease. Mitochondrial function will also studied.

1. The investigators hypothesize that both structure of sarcolemma and localization of key Ca2+-handling proteins are altered in patients with atrial fibrillation compared with patients in sinus rhythm.
2. The investigators hypothesize that mitochondrial function is altered in patients with atrial fibrillation compared with patients in sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* sinus rhythm, permanent atrial fibrillation or paroxysmal atrial fibrillation
* selected for open heart surgery
* informed consent

Exclusion Criteria:

* not given informed consent

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: selected for open heart surgery in St Olavs Hospital, Trondheim University Hospital, Norway
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
structure of sarcolemma | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, PhD, Study Director — Norwegian University of Science and Technology

REFERENCES:
- [Result] Slagsvold KH, Johnsen AB, Rognmo O, Hoydal MA, Wisloff U, Wahba A. Mitochondrial respiration and microRNA expression in right and left atrium of patients with atrial fibrillation. Physiol Genomics. 2014 Jul 15;46(14):505-11. doi: 10.1152/physiolgenomics.00042.2014. Epub 2014 May 13. PMID 24824214